CLINICAL TRIAL: NCT03523689
Title: Prevalence and Location of Intra-Procedural Atelectasis Detected by Radial-Probe Endobronchial Ultrasound During Peripheral Bronchoscopy Under General Anesthesia
Brief Title: Radial-Probe Endobronchial Ultrasound in Detecting Atelectasis in Patients Undergoing Peripheral Bronchoscopy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0123; NCI-2018-00964 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0123 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Malignant Neoplasms of Respiratory and Intrathoracic Organs; Lung Neoplasm
Keywords: Malignant neoplasms of respiratory and intrathoracic organs; Endobronchial ultrasound-guided transbronchial needle aspiration; EBUS-TBNA
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (bronchoscopy, RP-EBUS): Patients undergo bronchoscopy per standard of care, RP-EBUS of the left and right lungs during bronchoscopy procedure, and RP-imaging over 3-5 minutes at the end of the bronchoscopy procedure.
  Interventions: Procedure: Bronchoscopy; Procedure: Radial Probe Endobronchial Ultrasound

INTERVENTIONS:
Procedure: Bronchoscopy — Undergo bronchoscopy
Procedure: Radial Probe Endobronchial Ultrasound — Undergo RP-EBUS
  Other Names: Radial EBUS; Radial Endobronchial Ultrasound; Radial Probe EBUS; Radial-Probe Endobronchial Ultrasound; RP-EBUS

SUMMARY:
This trial studies how well radial-probe endobronchial ultrasound works in detecting the complete or partial collapse of the lung in patients undergoing peripheral bronchoscopy. Diagnostic procedures, such as radial-probe endobronchial ultrasound and bronchoscopy, use a thin, tube-like instrument inserted through the nose or mouth to view and take pictures of the inside of the trachea, air passages, and lungs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients identified as developing intraprocedural atelectasis detected by radial-probe endobronchial ultrasound (RP-EBUS) during peripheral bronchoscopy under general anesthesia.

SECONDARY OBJECTIVES:

I. To describe the most common locations for developing intraprocedural atelectasis detected by RP-EBUS.

II. To describe the proportion of evaluated bronchial segments per patient that are identified as developing intraprocedural atelectasis by RP-EBUS.

III. To identify patient and procedural characteristics that may predispose to the development of atelectasis.

OUTLINE:

Patients undergo bronchoscopy per standard of care, RP-EBUS of the left and right lungs during bronchoscopy procedure, and RP-imaging over 3-5 minutes at the end of the bronchoscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bronchoscopy with radial EBUS for peripheral lung lesions
* Recent computed tomography (CT) performed no more than 4 weeks prior to the bronchoscopy
* Voluntary informed consent to participate in the study

Exclusion Criteria:

* Patients with baseline lung consolidation, interstitial changes or lung masses (> 3 cm in diameter) in dependent areas of the lung as seen on most recent CT
* Pregnancy
* Ascites
* Known diaphragmatic paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing bronchoscopy with radial EBUS for peripheral lung lesions
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
New atelectasis for each segment | Up to 3 years
  Presence or absence of atelectasis within each of the aforementioned 8 segments will be determined using radial-probe endobronchial ultrasound (RP-EBUS) in comparison with the most recent computed tomography (CT) performed < 4 weeks prior to the bronchoscopy. A segment will be identified as having a new atelectasis if there is an indication of solid- or semisolid-appearing lesion by RP-EBUS without a corresponding indication of solid tumor or atelectasis on the preoperative CT. Descriptive statistics (frequencies, proportions, means, standard deviations, and ranges) will be provided for patient characteristics. The proportion of patients identified as developing intraprocedural atelectasis by RP-EBUS and its 95% confidence interval will be estimated to accomplish the primary objective.
Atelectasis for each patient | Up to 3 years
  Patients with at least 1 segment containing a new atelectasis will be determined to have atelectasis. Patients without atelectasis within any of the 8 segments will be determined to not have atelectasis. The proportion of patients identified as developing intraprocedural atelectasis by RP-EUS and its 95% confidence interval will be estimated to accomplish the primary objective.

SECONDARY OUTCOMES:
Common locations exhibiting atelectasis | Up to 3 years
  Locations of atelectasis will be summarized by a frequency table, allowing for multiple locations in the same patient.
Proportion of evaluated bronchial segments developing intraprocedural atelectasis | Up to 3 years
  The proportion of segments identified as developing atelectasis among all evaluated segments will be calculated for each patient, and the distribution of the proportion will be summarized by the mean, median, and range. We will compare patients with atelectasis and patients without atelectasis in terms of patient characteristics using a t-test or Wilcoxon test for continuous variables and Fisher's exact test or chi-squared test for categorical variables.
Patient characteristics associated with the presence of atelectasis | Up to 3 years
  To identify patient characteristics associated with the presence of atelectasis, logistic regression analysis will be used if the number of patients with atelectasis is at least 10. Due to a small sample size, multivariate logistic regression analysis may not be applied. A p-value of less than 0.05 will indicate statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Casal, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Sagar AS, Sabath BF, Eapen GA, Song J, Marcoux M, Sarkiss M, Arain MH, Grosu HB, Ost DE, Jimenez CA, Casal RF. Incidence and Location of Atelectasis Developed During Bronchoscopy Under General Anesthesia: The I-LOCATE Trial. Chest. 2020 Dec;158(6):2658-2666. doi: 10.1016/j.chest.2020.05.565. Epub 2020 Jun 17. PMID 32561439
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org